CLINICAL TRIAL: NCT00199875
Title: Cohort Study of Increasing Doses of Yttrium-90 Conjugated to Chimeric Monoclonal Antibody cG250 (^90Y-DOTA-cG250) in Patients With Advanced Renal Cancer
Brief Title: Treatment of Patients With Advanced Renal Cancer With a Radiolabeled Antibody, Yttrium-90 Conjugated Chimeric G250
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LUD2002-022; MSKCC IRB #: 05-031 (Other: MSKCC IRB)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2018-11-28 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Renal Cell Carcinoma; Kidney Neoplasm; Renal Cancer; Kidney Cancer
Keywords: antibody; renal cell carcinoma; advanced renal cancer; cG250; ^90Y
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients were enrolled sequentially in cohorts of 3 to 6 patients to receive escalating doses of study treatment until determination of the MTD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (0.2 mCi/kg) (Experimental): Patients initially received a nontherapeutic injection of ^111In-DOTA-cG250 (5 mCi ^111In + 10 mg cG250) on Day 1. Pending satisfaction of protocol-specified lesion targeting criteria, a single dose of therapeutic ^90Y-DOTA-cG250 (0.2 mCi/kg ^90Y + 10 mg cG250) was administered on Day 8, 9, or 10 as a continuous IV infusion over approximately 5 to 15 minutes.
  Interventions: Drug: Yttrium-90 conjugated chimeric G250 (^90Y-DOTA-cG250)
- Cohort 2 (0.3 mCi/kg) (Experimental): Patients initially received a nontherapeutic injection of ^111In-DOTA-cG250 (5 mCi ^111In + 10 mg cG250) on Day 1. Pending satisfaction of protocol-specified lesion targeting criteria, a single dose of therapeutic ^90Y-DOTA-cG250 (0.3 mCi/kg ^90Y + 10 mg cG250) was administered on Day 8, 9, or 10 as a continuous IV infusion over approximately 5 to 15 minutes.
  Interventions: Drug: Yttrium-90 conjugated chimeric G250 (^90Y-DOTA-cG250)
- Cohort 3 (0.4 mCi/kg) (Experimental): Patients initially received a nontherapeutic injection of ^111In-DOTA-cG250 (5 mCi ^111In + 10 mg cG250) on Day 1. Pending satisfaction of protocol-specified lesion targeting criteria, a single dose of therapeutic ^90Y-DOTA-cG250 (0.4 mCi/kg ^90Y + 10 mg cG250) was administered on Day 8, 9, or 10 as a continuous IV infusion over approximately 5 to 15 minutes.
  Interventions: Drug: Yttrium-90 conjugated chimeric G250 (^90Y-DOTA-cG250)
- Cohort 4 (0.45 mCi/kg) (Experimental): Patients initially received a nontherapeutic injection of ^111In-DOTA-cG250 (5 mCi ^111In + 10 mg cG250) on Day 1. Pending satisfaction of protocol-specified lesion targeting criteria, a single dose of therapeutic ^90Y-DOTA-cG250 (0.45 mCi/kg ^90Y + 10 mg cG250) was administered on Day 8, 9, or 10 as a continuous IV infusion over approximately 5 to 15 minutes.
  Interventions: Drug: Yttrium-90 conjugated chimeric G250 (^90Y-DOTA-cG250)
- Cohort 5 (0.55 mCi/kg) (Experimental): Patients initially received a nontherapeutic injection of ^111In-DOTA-cG250 (5 mCi ^111In + 10 mg cG250) on Day 1. Pending satisfaction of protocol-specified lesion targeting criteria, a single dose of therapeutic ^90Y-DOTA-cG250 (0.55 mCi/kg ^90Y + 10 mg cG250) was administered on Day 8, 9, or 10 as a continuous IV infusion over approximately 5 to 15 minutes.
  Interventions: Drug: Yttrium-90 conjugated chimeric G250 (^90Y-DOTA-cG250)

INTERVENTIONS:
Drug: Yttrium-90 conjugated chimeric G250 (^90Y-DOTA-cG250) — Patients received a single infusion of ^90Y-DOTA-cG250, with escalating doses administered to sequentially enrolled cohorts until MTD determination.

SUMMARY:
This was a Phase 1, open-label, dose-escalation study of yttrium-90 conjugated chimeric G250 (^90Y-DOTA-cG250) in patients with advanced, measurable clear cell renal cell carcinoma (RCC). Study objectives were to determine the safety, targeting, and dosimetry of ^90Y-DOTA-cG250, using indium-111 conjugated chimeric G250 (^111In-DOTA-cG250) as a surrogate, as well as to evaluate the immunogenicity of cG250.

DETAILED DESCRIPTION:
Patients were enrolled sequentially into cohorts of 3 to 6 patients until determination of the maximum tolerated dose (MTD) of ^90Y-DOTA-cG250, defined as the dose level below the dose at which ≥ 2 patients experienced dose-limiting toxicity (DLT). In an attempt to mitigate liver uptake and toxicity, patients initially received a nontherapeutic injection with ^111In-DOTA-cG250 at an imaging dose of 5 mCi of ^111In + 10 mg of cG250 on Day 1. Whole body and blood measurements of radioactivity were obtained on at least 3 occasions for 1 week to determine targeting and dosimetry. Provided that protocol-specified criteria were met, including targeting to lesions > 2 cm detected on computed tomography (CT) scan, a single dose of therapeutic ^90Y-DOTA-cG250 was administered on Day 8, 9, or 10. The starting dose of ^90Y-DOTA-cG250 was 0.2 mCi/kg of ^90Y + 10 mg of cG250 administered as an intravenous (IV) infusion, with escalation of the ^90Y dose in subsequent cohorts in 0.05 to 0.1 mCi/kg increments.

Patients were treated in an outpatient setting and were observed for at least 2 hours following each infusion, at which point vital signs and blood samples were obtained. Patients were followed for 6 to 8 weeks post-treatment (or after recovery from toxicity) with imaging, biochemical, serological, and hematologic tests to determine the safety of ^90Y-DOTA-cG250 and to inform dose-escalation decisions. Extent of disease evaluations, preferably by positron emission tomography (PET)/CT or standard CT, were performed at baseline and 6 to 8 weeks post-treatment (or after recovery from toxicity). Long-term follow-up was performed, when possible, every 12 weeks thereafter for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have had histologically proven clear cell renal carcinoma.
2. Age ≥ 18 years. Children were not enrolled because clear cell renal cancer is rarely seen in children.
3. All patients must have had a clinical presentation consistent with metastatic renal carcinoma.
4. Patients must have had bidimensionally measurable disease by conventional imaging methods including radiography, ultrasound, CT, or other anatomic imaging modalities. Lesions seen on skeletal scintigraphy alone were not considered measurable.
5. Female patients of childbearing age were required to have a negative pregnancy test carried out the day of and prior to receiving therapy, and were asked to use effective contraception during the study.
6. All patients must have been ambulatory with a Karnofsky Performance Status of at least 70.
7. The following laboratory results within the last 2 weeks prior to study Day 1:

   * serum creatinine ≤ 2.0 mg/dL
   * serum bilirubin (total) ≤ 2.0 mg/dL
   * aspartate aminotransferase (AST) ≤ 2.5 × the upper limit of normal (ULN)
   * alanine aminotransferase (ALT) ≤ 2.5 × ULN
   * white blood cell (WBC) count ≥ 3500/mm^3
   * platelet count ≥ 100,000/mm^3
   * prothrombin time ≤ 1.3 × control
8. Able and willing to give valid written informed consent.

Exclusion Criteria:

1. Significant prior radiotherapy (> 30 Gy) to the entire pelvis and/or lumbosacral spine.
2. Clinically significant cardiac disease (New York Heart Association Class [III/IV]).
3. Serious infection requiring treatment with antibiotics, or other serious illness.
4. Chemotherapy, radiation therapy, or immunotherapy within 4 weeks prior to study agent administration.
5. Survival expectancy of less than 12 weeks.
6. Patients with central nervous system (CNS) involvement were excluded under the following criteria:

   * Brain metastasis, except for stable disease over 3 months.
   * Untreated brain metastasis.
   * Evidence of progression of neurologic CNS involvement within 3 months prior to entering the protocol.
7. Hypercalcemia > 12.5 mg/100 mL or symptomatic.
8. Mental impairment that may have compromised the ability to give informed consent and comply with the requirements of the study.
9. Lack of availability of the patient for clinical and laboratory follow-up assessment.
10. Patients known to have hepatobiliary disease and/or human immunodeficiency virus/acquired immune deficiency syndrome.
11. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.
12. Pregnancy or breastfeeding.
13. Refusal or inability to use effective means of contraception in men or women of childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-07-06 (Actual); Primary Completion 2013-03-14 (Actual); Study Completion 2013-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Larson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Neeta Pandit-Taskar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Joseph O'Donoghue, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Robert Motzer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 (0.2 mCi/kg) | Cohort 2 (0.3 mCi/kg) | Cohort 3 (0.4 mCi/kg) | Cohort 4 (0.45 mCi/kg) | Cohort 5 (0.55 mCi/kg)
Started | 3 | 3 | 6 | 3 | 3
Completed | 3 | 3 | 6 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set includes all patients who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (0.2 mCi/kg) | Cohort 2 (0.3 mCi/kg) | Cohort 3 (0.4 mCi/kg) | Cohort 4 (0.45 mCi/kg) | Cohort 5 (0.55 mCi/kg) | Total
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 3 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (9.2) | 64.7 (4.9) | 62.7 (7.9) | 63.7 (6.8) | 63.0 (5.9) | 63.7 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 0 | 2 | 7
  Male | 2 | 2 | 3 | 3 | 1 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6 | 3 | 3 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1
  White | 3 | 3 | 6 | 2 | 2 | 16
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6 | 3 | 3 | 18
Karnofsky Performance Status [Count of Participants; unit: Participants] — Higher performance status indicates higher functional abilities, as follows:
  100=Normal, no complaints/evidence of disease. 90=Able to carry on normal activity; minor signs/symptoms of disease. 80=Normal activity with effort; some signs/symptoms of disease. 70=Cares for self; unable to carry on normal activity or do active work. 60=Requires occasional assistance but is able to care for most personal needs. 50=Requires considerable assistance & frequent medical care. 0-40=Unable to care for self; requires equivalent of institutional or hospital care; disease may be progressing rapidly.
  Participants
    70 | 0 | 0 | 1 | 0 | 0 | 1
    80 | 1 | 0 | 1 | 0 | 3 | 5
    90 | 2 | 2 | 3 | 2 | 0 | 9
    100 | 0 | 0 | 1 | 1 | 0 | 2
    Missing | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment-emergent Adverse Events
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Toxicity Criteria (CTC), version 3.0. Treatment-emergent adverse events (TEAEs) were reported based on clinical laboratory tests, physical examinations, and vital signs from pre-treatment through the study period. Dose-limiting toxicity (DLT) was defined as follows for the purposes of dose escalation: Grade 4 hematopoietic toxicity in excess of 5 days or Grade 3 or greater nonhematopoietic toxicity.
Time Frame: Continuously for up to 5 months
Population: The Safety Analysis Set includes all patients who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (0.2 mCi/kg) | Cohort 2 (0.3 mCi/kg) | Cohort 3 (0.4 mCi/kg) | Cohort 4 (0.45 mCi/kg) | Cohort 5 (0.55 mCi/kg)
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 3
Participants
  Any TEAE | 3 | 3 | 6 | 3 | 3
  Maximum grade 1 TEAE | 2 | 2 | 2 | 1 | 0
  Maximum grade 2 TEAE | 0 | 1 | 1 | 0 | 0
  Maximum grade 3 TEAE | 1 | 0 | 3 | 1 | 1
  Maximum grade 4 TEAE | 0 | 0 | 0 | 1 | 2
  Treatment-related TEAE | 2 | 3 | 5 | 3 | 3
  Serious TEAE | 0 | 0 | 1 | 1 | 0
  TEAE Leading to Treatment Discontinuation | 0 | 0 | 0 | 0 | 0
  TEAE Meeting DLT Criteria | 0 | 0 | 1 | 0 | 2

2. Secondary Outcome: Number of Patients Who Met Protocol-Specified Criteria to Receive ^90-Y-DOTA-cG250 Following ^111In-DOTA-cG250 Administration
Description: In order to receive the therapeutic ^90Y-DOTA-cG250 injection on Day 8, 9, or 10, patients must have demonstrated tumor targeting to lesions > 2 cm detected by CT scan and must not have exhibited the following characteristics following the nontherapeutic injection of ^111In-DOTA-cG250: excessive liver and/or spleen uptake; excessive uptake in the normal kidney; non-visualization of the cardiac blood pool in the first imaging set; whole body clearance half-life (t1/2) < 1.5 days; serum t1/2 < 2 days; rapid clearance of the radiopharmaceutical from the blood pool with prominent marrow uptake on the first image.
Time Frame: Up to 5 months
Population: The Safety Analysis Set includes all patients who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (0.2 mCi/kg) | Cohort 2 (0.3 mCi/kg) | Cohort 3 (0.4 mCi/kg) | Cohort 4 (0.45 mCi/kg) | Cohort 5 (0.55 mCi/kg)
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 3
Participants | 3 | 3 | 6 | 3 | 3

3. Secondary Outcome: Number of Patients With Samples Collected for Evaluation of Human Antichimeric Antibody
Description: Blood samples were drawn for evaluation of the human antichimeric antibody (HACA) at screening, between Days 22 and 28, between Days 36 and 42, between Days 43 and 57 or at the end of study, and during long-term follow-up (approximately 12 weeks later). Serial dilutions were tested by the enzyme-linked immunosorbent assay (ELISA) using the "double antibody sandwich" technique and pretreatment serum as negative control.
Time Frame: Up to 6 months
Population: The Safety Analysis Set includes all patients who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (0.2 mCi/kg) | Cohort 2 (0.3 mCi/kg) | Cohort 3 (0.4 mCi/kg) | Cohort 4 (0.45 mCi/kg) | Cohort 5 (0.55 mCi/kg)
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 3
Participants
  Baseline | 3 | 3 | 6 | 3 | 3
  Day 28 | 3 | 3 | 6 | 3 | 3
  Day 42 | 3 | 3 | 6 | 3 | 3
  Day 63 | 3 | 3 | 6 | 2 | 2
  Long-term Follow-up | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring between the signing of informed consent and the off-study date were documented, regardless of the causal relationship to study drug. AEs occurring after the first dose of study drug were considered treatment emergent (i.e., TEAEs). The AE reporting period for this study was up to 5 months.
Description: AE documentation included onset/resolution dates, severity using the NCI CTC (version 3.0), seriousness, study drug action taken, treatment, and outcome. In summaries, treatment-related AEs included those with a "possible", "probable", or "definite" relationship to study drug; preferred terms were counted only once per patient at the maximum reported grade.
Arm/Group | Cohort 1 (0.2 mCi/kg) | Cohort 2 (0.3 mCi/kg) | Cohort 3 (0.4 mCi/kg) | Cohort 4 (0.45 mCi/kg) | Cohort 5 (0.55 mCi/kg)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/6 | 1/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (0.2 mCi/kg) (N=3) | Cohort 2 (0.3 mCi/kg) (N=3) | Cohort 3 (0.4 mCi/kg) (N=6) | Cohort 4 (0.45 mCi/kg) (N=3) | Cohort 5 (0.55 mCi/kg) (N=3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (0.2 mCi/kg) (N=3) | Cohort 2 (0.3 mCi/kg) (N=3) | Cohort 3 (0.4 mCi/kg) (N=6) | Cohort 4 (0.45 mCi/kg) (N=3) | Cohort 5 (0.55 mCi/kg) (N=3)
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase (Investigations) | 2 | 0 | 3 | 1 | 1
Haemoglobin (Investigations) | 2 | 0 | 5 | 3 | 3
International normalised ratio (Investigations) | 2 | 0 | 1 | 1 | 1
Platelet count (Investigations) | 2 | 3 | 5 | 3 | 3
Alanine aminotransferase (Investigations) | 1 | 0 | 1 | 0 | 2
Blood creatinine (Investigations) | 1 | 2 | 5 | 1 | 1
Prothrombin time (Investigations) | 1 | 0 | 1 | 0 | 1
White blood cell count (Investigations) | 1 | 2 | 3 | 2 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 3 | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 6 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Amylase (Investigations) | 0 | 1 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 3
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 1 | 3
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase (Investigations) | 0 | 0 | 2 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Neutrophil count (Investigations) | 0 | 0 | 1 | 0 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less